CLINICAL TRIAL: NCT06147570
Title: A Phase II, Open-label, Multicenter Study to Evaluate the Efficacy，Safety and Pharmacokinetics of HS-10365 as First-Line Treatment for Patients With Locally Advanced or Metastatic RET Fusion-Positive Non-Small Cell Lung Cancer
Brief Title: A Study of HS-10365 in Patients With Advanced or Metastatic RET Fusion-Positive Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10365-201
Record Dates: First submitted 2023-11-17; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10365 (Experimental): 160 mg BID of HS-10365
  Interventions: Drug: HS-10365 capsules

INTERVENTIONS:
Drug: HS-10365 capsules — HS-10365 will be administered orally twice daily until the occurrence of disease progression, unacceptable adverse events, withdrawal of consent, death or the end of the study.

SUMMARY:
HS-10365 is a small molecular, oral potent, selective RET inhibitor. The purpose of this study is to investigate the efficacy and safety of HS-10365 in Chinese advanced RET fusion-positive non-small cell lung cancer patients without any systemic therapy.

DETAILED DESCRIPTION:
This is an open-label, single arm, multi-center Phase 2 study in participants with treatment-naïve locally advanced or metastatic RET fusion-positive non-small cell lung cancer, which is designed to investigate the anti-tumor activity, safety and pharmacokinetics (PK) of HS-10365 at the recommended phase 2 dose (RP2D). HS-10365 will be administered orally twice daily until the occurrence of disease progression, unacceptable adverse events, withdrawal of consent, death or the end of the study. Primary endpoint is objective response rate (ORR) by Independent Reading Committee (IRC). Secondary and exploratory objectives include evaluation of secondary efficacy endpoints, safety and PK in the study population.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged more than or equal to (≥) 18 years.
2. Histologically or cytologically confirmed diagnosis of locally advanced or metastatic NSCLC with RET fusion-positive, including recurrent or initial diagnosed Stage IIIB-IIIC/IV NSCLC that is not suitable for radical surgery.
3. A RET gene fusion is required by using tumor tissue for central testing.
4. At least one measurable lesion in accordance with RECIST 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status: 0~1.
6. Estimated life expectancy >12 weeks.
7. Reproductive-age women agree to use adequate contraception and cannot breastfeed while participating in this study and for a period of 6 months after the last dose. Likewise, men also consent to use adequate contraceptive method within the same time limit.
8. Females must have evidence of non-childbearing potential.
9. Signed and dated Informed Consent Form.

Exclusion Criteria:

1. Treatment with any of the following:

   Additional validated oncogenic drivers in NSCLC if known. Previous or current treatment with selective RET inhibitors or multi-kinase Inhibitor of RET.

   Prior systemic therapy for metastatic disease. Treatment (including chemotherapy or immunotherapy) in the adjuvant/neoadjuvant setting is permitted if it was completed at least 6 months prior to relapse.

   Local radiotherapy for palliation within 2 weeks of the first dose of study drug, or patients received more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks of the first dose.

   Major surgery (including craniotomy, thoracotomy, or laparotomy, etc.) within 4 weeks of the first dose of study drug.
2. Inadequate bone marrow reserve or serious organ dysfunction.
3. Uncontrolled pleural effusion or ascites or pericardial effusion.
4. Known and untreated, or active central nervous system metastases.
5. Active autoimmune diseases or active infectious disease
6. Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow oral medications.
7. History of severe allergic reaction, hypersensitivity to any active or inactive ingredient of HS-10365 or to drugs with a similar chemical structure or class to HS-10365.
8. The subject who is unlikely to comply with study procedures, restrictions, or requirements judged by the investigator.
9. The subject whose safety cannot be ensured or study assessments would be interfered judged by the investigator.
10. Pregnant women, breastfeeding women or woman who has a child-bearing plan during the study.
11. History of neuropathy or mental disorders, including epilepsy and dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
ORR assessed by IRC | From the date of first occurrence of complete response (CR) or partial response (PR) on 2 consecutive occasions (≥4 weeks), until the date of disease progression or withdrawal from study, whichever came first, up to 48 months.
  ORR is defined as the percentage of patients with a CR or PR that was confirmed at a subsequent scan at least 4 weeks later, as assessed according to RECIST version 1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | From the first occurrence of confirmed CR or PR or SD until the date of disease progression or withdrawal from study, whichever came first, up to 48 months.
  Objective response was assessed by RECIST 1.1 thereby to evaluate disease control rate. Disease control was deﬁned as the percentage of patients who have a best overall response (confirmed CR, PR, or stable disease for at least 5 weeks).
Duration of response (DOR) | From the date of the first dose to disease progression or death in patients who achieve CR or PR, whichever came first, up to 48months.
  Duration of response (DOR)
Progression-free survival (PFS) | From the date of the first dose until the date of disease progression or death from any cause, whichever came first, up to 48 months.
  Progression of tumor was assessed by RECIST 1.1 thereby to evaluate progression free survival. Progression-free survival was deﬁned as the time from date of ﬁrst dose until the documentation of objective PD or death from any cause in the absence of progression (whichever occurred first), regardless of whether they subsequently received non-study anti-cancer therapy.
Overall survival (OS) | The time from initial administration to death from any cause, up to 5 years.
  Overall survival (OS)
Incidence and severity of treatment-related adverse events | From the first dose until 28 days after the last dose
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, and NCI CTCAE v5.0.
Observed maximum plasma concentration (Cmax) of HS-10365 | At the firs of every Cycle from 1 to 12（each cycle is 28 days）
  Cmax of HS-10365

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided